CLINICAL TRIAL: NCT02105792
Title: PROspective Cohort MRC ABPI STratification and Extreme Response Mechanism in Diabetes
Brief Title: PROMASTER - PROspective Cohort MRC ABPI STratification and Extreme Response Mechanism in Diabetes
Acronym: PROMASTER
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); King's College London (Other); King's College Hospital NHS Trust (Other); University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other); Newcastle University (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRF112; 12/SW/0347 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Diabetes
Keywords: Diabetes; Type 2 diabetes; Diabetes therapy response; Diabetes progression
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Sulfonylurea Compounds; Dipeptidyl-Peptidase IV Inhibitors; Sodium-Glucose Transporter 2 Inhibitors; Thiazolidinediones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At Visit 1, a fasting blood sample (approximately 35 ml) will be collected for DNA extraction, and to measure for markers of the progression of diabetes or response to diabetes medication and for secondary markers that may predict response. A urine sample is also collected to measure for biomarkers.
  At Visit 2 a fasting blood sample and urine sample will be collected to measure for markers of the response to diabetes medication and for secondary markers that may predict response.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Responders: Patients with Type 2 diabetes about to commence a second- or third-line glucose-lowering treatment (Sulphonylurea, DPP-4 inhibitors, GLP-1R agonists, SGLT2 inhibitors or Glitazone or insulin).
  Interventions: Drug: second- or third-line glucose-lowering diabetes treatment
- Progressors: Patients with Type 2 diabetes that progress to requiring insulin treatment ≤10 years from diagnosis or have no requirement for insulin treatment >10 years from diagnosis.

INTERVENTIONS:
Drug: second- or third-line glucose-lowering diabetes treatment — Observation of response and disease progression following clinician's addition of a glucose-lowering diabetes therapy (Sulphonylurea, DPP-4 inhibitor, GLP-1R agonist, SGLT2 inhibitor or Glitazone) to existing therapy.
  Other Names: Sulphonylurea; DPP-4 inhibitor; GLP-1R agonist; SGLT2 inhibitor; Glitazone
  Groups: Responders

SUMMARY:
This study will examine extreme responders to second- and third-line Type 2 diabetes therapy using a prospective approach, and patients with slow or fast diabetes progression using a retrospective approach.

DETAILED DESCRIPTION:
PILOT Phase (March 2013 - Dec 2014) Participants will be recruited initially from 4 centres. Patients due to start second- and third-line Type 2 diabetes treatments, and patients progressing to insulin either particularly quickly or particularly slowly, will be recruited from primary care, secondary care, or community settings. Fasting blood and urine samples will be collected, together with standard biomeasures and information about medical history and prescribing history. Participants in Responders Arm will be contacted by telephone approximately 3 months after starting their new second/third-line agent to review their current medication and blood glucose level. If a 3 month HbA1c has not been collected as part of routine clinical care, the research team will arrange this. Participants will be asked to return for a blood and urine test approximately 6 months after their new treatment was started. This visit will be brought forward should the participant advise they are about to further change their treatment, to enable their samples to be collected in advance of their proposed treatment change.

All study documentation and sample materials will be distributed to sites from the Coordinating Centre. Sites will be expected to process and freeze samples and send them to the Chief Investigator's Central Laboratory where they will be analysed for genetic factors, glycaemic markers and other markers related to drug response.

POST-PILOT Phase (Jan 2015 - Oct 2017) Subject to feasibility, interim analysis and continuation of funding from Medical Research Council (MRC), this study will continue for another 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: Age 18-90 inclusive
* Ethnicity: Reflective of local demographic
* Medical History: Clinical diagnosis of Type 2 diabetes
* Mental Capacity: Capacity to Consent

Exclusion Criteria:

* Age less than 18 years old and greater than 90 years old
* Incapacity to consent
* Type 1 diabetes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified in primary care and secondary care. The method for patient identification may differ between sites and could involve:
  GP Searches; Secondary Care Clinician Referral; Research Database Searches.
Sampling Method: Non-Probability Sample
Enrollment: 820 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Response to diabetes therapy | Up to 9 months from commencement of new therapy
  The primary outcome will be to compare the clinical characteristics of the patients who show an excellent response or a poor response to specific second- and third-line classes of treatment for Type 2 diabetes.

SECONDARY OUTCOMES:
Collection of samples for analysis of potential biomarkers | within 9 months of recruitment date
  To collect a set of DNA, serum and urine samples to allow analysis of potential genetic and non genetic biomarkers for drug response and diabetes progression.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, FRCP, DM, BM, Principal Investigator — University of Exeter
Locations (5):
- United Kingdom (5):
  - University of Exeter, Exeter, Devon
  - Oxford University Hospitals NHS Trust, Oxford, Oxfordshire
  - University of Newcastle, Newcastle upon Tyne, Tyne and Wear
  - University of Glasgow, Glasgow
  - King's College University of London, London

IPD SHARING:
Plan to Share IPD: No